CLINICAL TRIAL: NCT03779659
Title: Effectiveness of Synapse Transcutaneous Electronic Nerve Stimulation (TENS) Device in Reducing Pain Among Children 6-14 Years During Dental Treatments in a Randomized Cross-over Clinical Trial
Brief Title: Effectiveness of Synapse Transcutaneous Electronic Nerve Stimulation (TENS) During Dental Procedures Among Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Prior to IRB submission, Covid-19 related logistical and personnel issues led to the decision to not move forward with this research.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-37546
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Dental Fear; Anesthesia, Local; Pediatric Dentistry
Keywords: Electronic dental anesthesia; Transcutaneous Electronic Nerve Stimulation (TENS); Topical anesthesia; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Benzocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Synapse TENS device (Experimental): SYnapse TENS device will be used for alleviating pain through electrical stimulation. This is a battery powered device where an electrical current is applied intra-orally on the buccal and lingual sides using an intra-oral pad applicator. This device has been cleared for marketing by the Food and Drug Administration (FDA) and the prescribed electrical field falls almost a 10 factor level lower than routine pulp testing devices used in dentistry. The TENS device was previously tested in a pilot study with promising results. Chair side application and at-home use of the device by the patient was shown to drastically reduce pain and discomfort associated with orthodontic tooth movement.
  Interventions: Device: Synapse TENS device
- Topical anesthetic gel (Active Comparator): Topical anesthetic Gel is the active comparator in this study. The topical anesthesia (anesthetic gel) Centrix LolliCaine with 20% benzocaine in single package of 0.3 ml will be used. The amount of local anesthetic used will not exceed the maximum allowable dose, which will be calculated for each patient based on his/her age and weight prior to the dental procedure. This will be done based American Association of Pediatric Dentistry guidelines for the use of local anesthesia.
  Interventions: Drug: Topical anesthetic gel

INTERVENTIONS:
Device: Synapse TENS device — At the time of local anesthetic application the TENS device will be activated and placed on the buccal and lingual alveolar mucosa adjacent to the tooth receiving the restorative treatment using the pad applicator. The tip of the device with the electrodes are placed in a vertical up and down motion for approximately ten seconds. Following this, the level of pain and anxiety are measured using the Wong Baker Scale and Visual Analog Scale. The TENS device is used for achieving localized pain relief at the site of local anesthetic injection prior to injecting the anesthetic agent (such as lidocaine or articaine). Following this, once the clinician ensures that the patient is pain free then local anesthetic injection is given and following that the dental procedures are conducted.
  Other Names: ALEVE therapy
  Arms: Synapse TENS device
Drug: Topical anesthetic gel — The local anesthetic gel is typically used for achieving localized pain relief at the site of local anesthetic injection and this is part of standard care that is followed prior to dental procedures.
  The amount of local anesthetic used will not exceed the maximum allowable dose, which will be calculated for each patient based on his/her age and weight prior to the dental procedure
  Other Names: Centrix LolliCaine 2% xylocaine with 20% benzocaine
  Arms: Topical anesthetic gel

SUMMARY:
Dental Fear and Anxiety (DFA) are at higher levels among children and often leads to avoidance of dental treatment. Negative experiences in the early years such as experience of pain during injections, fillings, or extractions may lead to difficulties in treatment and behavior management among children. During dental procedures such as restorations and extractions injectable anesthetics are required as they are used to anesthetize and numb the area around the tooth receiving treatment. Topical anesthetics are used prior to using injectable anesthetic to alleviate some pain and discomfort. Topical anesthetics should be used with caution as they consist of more concentrated doses of pharmaceutical elements used in injectable anesthetics. Such high concentrations can result in increased gag reflux, central nervous system depression and cardiovascular effects in rare cases. With many recent advances in dental treatment, there is also a need for new non-pharmaceutical strategies to alleviate pain and discomfort among children which in turn will motivate children and their parents to visit the dental clinic more frequently. Electronic anesthesia or Synapse Transcutaneous Electronic Nerve Stimulation (TENS), a non-invasive device that uses low energy electrical stimulation to reduce pain perception, has gained acceptance since the 1990s. Advantages of using the TENS device are that it is safe, easy to use, well-accepted among patients as evidenced in the few trials conducted so far, no adverse complications and has been successful in alleviating pain during dental procedures. This study aims to explore use of the TENS to alleviate pain and discomfort at the oral mucosal site where the patient will receive a local anesthetic injection. In this randomized case-crossover trial among children aged 6-14 years the effectiveness of Aleve TENS device in reducing pain and anxiety among children prior to receiving injectable local anesthetic agent during dental procedures is compared to those who receive the local anesthetic gel prior to receiving local anesthetic injection.

DETAILED DESCRIPTION:
Children between 6-14 years will be recruited at the Pediatric Oral Healthcare Center. A sample of 100 male and female children who fit the inclusion and exclusion criteria are recruited. Once parents' consent at the first visit basic demographic information, dental and medical history information is collected. This study is conducted in total of two clinic visits. In the first visit participants are randomized to either the intervention group or the comparison group. The intervention group receives the experimental device (TENS) prior to local anesthetic injection whereas the comparison group receives the local anesthetic gel. Following this the participants receive the local anesthetic injection after which treatment is completed. In the second visit the participants are crossed over to the other group and therefore randomization is not used for visit 2. Those who received the local anesthetic gel in visit 1 will receive the experimental device in visit 2 and those who received the experimental device in visit 1 will receive the local anesthetic gel in visit 2 . Following this treatment procedures are completed.

ELIGIBILITY:
Inclusion Criteria:

* Children who are healthy and without any major medical conditions
* Children who are patients at the Pediatric Oral Healthcare Center
* Children requiring restoration on the occlusal surface that involves tooth preparation up to the dentin level in at least two primary or permanent molars or children requiring extractions of primary or permanent molars.
* Children who are scheduled for at least two appointments and who require two restorative procedures or two extractions than can be scheduled over two separate appointments

Exclusion Criteria:

* Children who have contraindications to local anesthetic
* Children with teeth requiring restoration and have pulp involvement and root resorption on radiological examination (i.e. deep caries)
* Children who have major medical problems
* Children taking medications for major medical illnesses
* Children who have pacemakers
* Children with ADD/ADHD, autism or Down's syndrome and children with a history of behavioral issues that required previous management.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Presence of Pain before treatment | before the start of each treatment procedure up to 6 months
  The presence of pain will be a simple question in the case report form with two answer choices: yes or no.
Presence of Pain before local analgesic injection | after TENS or gel administration before local analgesic injection at about 1 minute
  The presence of pain will be a simple question in the case report form with two answer choices: yes or no.
Presence of Pain after treatment | about 45 minutes at the end of the treatment visit
  The presence of pain will be a simple question in the case report form with two answer choices: yes or no.
Level of pain before treatment based on Wong-Baker Faces (WBF) pain rating scale | before the start of each treatment procedure up to 6 months
  Level of pain will be measured using the Wong-Baker Faces (WBF) pain rating scale. The scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value from 0 to 5, with higher values indicating more pain. Based on child's selection of the facial expression a score will be assigned.
Level of pain before local analgesic injection based on Wong-Baker Faces (WBF) pain rating scale | after TENS or gel administration before local analgesic injection at about 1 minute
  Level of pain will be measured using the Wong-Baker Faces (WBF) pain rating scale. The scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value from 0 to 5, with higher values indicating more pain. Based on child's selection of the facial expression a score will be assigned.
Level of pain after treatment based on Wong-Baker Faces (WBF) pain rating scale | about 45 minutes at the end of the treatment visit
  Level of pain will be measured using the Wong-Baker Faces (WBF) pain rating scale. The scale is a set of six cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Each face has a numeric value from 0 to 5, with higher values indicating more pain. Based on child's selection of the facial expression a score will be assigned.
Level of dental anxiety before treatment using Visual Analog Scale | before the start of each treatment procedure up to 6 months
  Level of anxiety will be measured using the Visual Analog Scale. The scale is a simple line with the number line ranging from 0 to 10. Children are asked how nervous or confident they feel and are asked to point or mark on the line. The corresponding numerical value will be noted for each patient.
Level of dental anxiety before local analgesic injection using Visual Analog Scale | after TENS or gel administration before local analgesic injection at about 1 minute
  Level of anxiety will be measured using the Visual Analog Scale. The scale is a simple line with the number line ranging from 0 to 10. Children are asked how nervous or confident they feel and are asked to point or mark on the line. The corresponding numerical value will be noted for each patient.
Level of dental anxiety after treatment using Visual Analog Scale | about 45 minutes at the end of the treatment visit
  Level of anxiety will be measured using the Visual Analog Scale. The scale is a simple line with the number line ranging from 0 to 10. Children are asked how nervous or confident they feel and are asked to point or mark on the line. The corresponding numerical value will be noted for each patient.

SECONDARY OUTCOMES:
Patient's comfort level preference | up to 6 months
  The comfort or preference level for TENS device versus local anesthetic gel prior to local anesthetic injection will be assessed by asking the participants about their preference using a question in the case report form with five answer choices (using Likert scale - Very uncomfortable, somewhat uncomfortable, neither comfortable nor uncomfortable, somewhat comfortable, very comfortable)..
Treatment completion status | up to 6 months
  Treatment completion status will be recorded as 'completed' or 'partially completed' on the Case Report Form at the conclusion of each treatment visit.
Reason for partially completed treatment | up to 6 months
  For participants that do not complete both treatment procedures and are categorized as 'incomplete', the reason/s why will be documented.
Supplemental anesthetic use | up to 6 months
  Amount of supplemental anesthesia if used for each of the two treatment procedures will be recorded in clinic notes after each treatment procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jayapriyaa Shanmugham, BDS DrPH, Principal Investigator — Department of Pediatric Dentistry, Henry M. Goldman School of Dental Medicine
Locations (1):
- BU Henry M. Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Overall findings and summary of results for primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Once data collection is complete and data analysis has been completed the results will be made available.
Access Criteria: Since this is a pilot study only summary data will be provided.

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. 4th ed. Washington DC, American Psychiatric Press. 1994.
- [Background] Alvesalo I, Murtomaa H, Milgrom P, Honkanen A, Karjalainen M, Tay KM. The Dental Fear Survey Schedule: a study with Finnish children. Int J Paediatr Dent. 1993 Dec;3(4):193-8. doi: 10.1111/j.1365-263x.1993.tb00083.x. PMID 8142322
- [Background] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Background] Cianetti S, Lombardo G, Lupatelli E, Pagano S, Abraha I, Montedori A, Caruso S, Gatto R, De Giorgio S, Salvato R. Dental fear/anxiety among children and adolescents. A systematic review. Eur J Paediatr Dent. 2017 Jun;18(2):121-130. doi: 10.23804/ejpd.2017.18.02.07. PMID 28598183
- [Background] Ogle OE, Mahjoubi G. Local anesthesia: agents, techniques, and complications. Dent Clin North Am. 2012 Jan;56(1):133-48, ix. doi: 10.1016/j.cden.2011.08.003. PMID 22117947
- [Background] Armfield JM, Milgrom P. A clinician guide to patients afraid of dental injections and numbness. SAAD Dig. 2011 Jan;27:33-9. PMID 21323034
- [Background] Lee HS. Recent advances in topical anesthesia. J Dent Anesth Pain Med. 2016 Dec;16(4):237-244. doi: 10.17245/jdapm.2016.16.4.237. Epub 2016 Dec 31. PMID 28879311
- [Background] Boyce RA, Kirpalani T, Mohan N. Updates of Topical and Local Anesthesia Agents. Dent Clin North Am. 2016 Apr;60(2):445-71. doi: 10.1016/j.cden.2015.12.001. PMID 27040295
- [Background] Yap AU, Ho HC. Electronic and local anesthesia: a clinical comparison for operative procedures. Quintessence Int. 1996 Aug;27(8):549-53. PMID 9161258
- [Background] Abdulhameed SM, Feigal RJ, Rudney JD, Kajander KC. Effect of peripheral electrical stimulation on measures of tooth pain threshold and oral soft tissue comfort in children. Anesth Prog. 1989 Mar-Apr;36(2):52-7. PMID 2604057
- [Background] teDuits E, Goepferd S, Donly K, Pinkham J, Jakobsen J. The effectiveness of electronic dental anesthesia in children. Pediatr Dent. 1993 May-Jun;15(3):191-6. PMID 8378157
- [Background] Cho SY, Drummond BK, Anderson MH, Williams S. Effectiveness of electronic dental anesthesia for restorative care in children. Pediatr Dent. 1998 Mar-Apr;20(2):105-11. PMID 9566014
- [Background] Baghdadi ZD. Evaluation of electronic dental anesthesia in children. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Oct;88(4):418-23. doi: 10.1016/s1079-2104(99)70055-7. PMID 10519748
- [Background] Oztas N, Olmez A, Yel B. Clinical evaluation of transcutaneous electronic nerve stimulation for pain control during tooth preparation. Quintessence Int. 1997 Sep;28(9):603-8. PMID 9477875
- [Background] Dhindsa A, Pandit IK, Srivastava N, Gugnani N. Comparative evaluation of the effectiveness of electronic dental anesthesia with 2% lignocaine in various minor pediatric dental procedures: A clinical study. Contemp Clin Dent. 2011 Jan;2(1):27-30. doi: 10.4103/0976-237X.79305. PMID 22114450